CLINICAL TRIAL: NCT03141138
Title: A Phase 1, Randomized, Open-label, Comparison of Heterologous Prime-Boost Vaccination Schedules of Tetravalent Dengue Virus Purified Inactivated Vaccine (PIV) and Tetravalent Dengue Virus Live Attenuated Vaccine (LAV) in Healthy Adults
Brief Title: Comparison of Tetravalent Dengue Virus Purified Inactivated Vaccine and Tetravalent Dengue Virus Live Attenuated Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-16-23
Record Dates: First submitted 2017-04-25; First posted 2017-05-04 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Dengue Virus

STUDY DESIGN:
Masking Description: This will be an open-label study. The laboratories in charge of testing will be blinded to the experimental arm, and codes will be used to link the subject and study (without any link to the experimental arm attributed to the subject) to each sample.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: TDENV-PIV on Day 0 (Experimental): Dosage: 0.5 mL of DENV serotypes 1-4 (4 µg / serotype) in alum adjuvant Mode of administration: intramuscular (IM) into the subject's upper arm, deltoid area of the subject's arm; vaccination will be given in the non-dominant arm whenever possible
  Interventions: Biological: TDENV-PIV
- Group 1: TDENV-LAV F17 on Day 180 (Experimental): Dosage: 0.5 mL of the post-transfection LAV F17 vaccine Mode of administration: subcutaneously into the upper-outer triceps/deltoid area of the subject's arm; vaccination will be given in the non-dominant arm whenever possible
  Interventions: Biological: TDENV-LAV F17
- Group 2: TDENV-PIV on Day 0 (Experimental): Dosage: 0.5 mL of DENV serotypes 1-4 (4 µg / serotype) in alum adjuvant Mode of administration: intramuscular (IM) into the subject's upper arm, deltoid area of the subject's arm; vaccination will be given in the non-dominant arm whenever possible
  Interventions: Biological: TDENV-PIV
- Group 2:TDENV-LAV F17 on Day 90 (Experimental): Dosage: 0.5 mL of the post-transfection LAV F17 vaccine Mode of administration: subcutaneously into the upper-outer triceps/deltoid area of the subject's arm; vaccination will be given in the non-dominant arm whenever possible
  Interventions: Biological: TDENV-LAV F17

INTERVENTIONS:
Biological: TDENV-PIV — Dosage: 0.5 mL of DENV serotypes 1-4 (4 µg / serotype) in alum adjuvant Mode of administration: intramuscular (IM) into the subject's upper arm, deltoid area of the subject's arm; vaccination will be given in the non-dominant arm whenever possible
  Arms: Group 1: TDENV-PIV on Day 0; Group 2: TDENV-PIV on Day 0
Biological: TDENV-LAV F17 — Dosage: 0.5 mL of the post-transfection LAV F17 vaccine Mode of administration: subcutaneously into the upper-outer triceps/deltoid area of the subject's arm; vaccination will be given in the non-dominant arm whenever possible.
  Arms: Group 1: TDENV-LAV F17 on Day 180; Group 2:TDENV-LAV F17 on Day 90

SUMMARY:
This study is a Phase 1, randomized, open-label study of the prime-boost vaccine candidates given in the prime-boost regimen previously demonstrated to have a high level of immunogenicity and immune durability: Day 0 prime (PIV) and Day 180 boost (LAV), and compare it with a previously untested schedule: Day 0 prime (PIV) and Day 90 boost (LAV) in order to define the potential tradeoff between potential immunogenicity, including cell-mediated immunity, and a more practical dosing schedule.

DETAILED DESCRIPTION:
This study is a Phase 1, randomized, open-label, study with 2 treatment groups (N=40):

Group 1 (n=20): TDENV-PIV 4 µg + Alum adjuvant (Day 0), TDENV-LAV F17 (Day 180) Group 2 (n=20): TDENV-PIV 4 µg + Alum adjuvant (Day 0), TDENV-LAV F17 (Day 90)

Investigational Product Dosage, Schedule, and Mode of Administration:

TDENV-PIV Dosage: 0.5 mL of DENV serotypes 1-4 (4 µg / serotype) in alum adjuvant Mode of administration: intramuscular (IM) into the subject's upper arm, deltoid area of the subject's arm; vaccination will be given in the non-dominant arm whenever possible TDENV-LAV F17 Dosage: 0.5 mL of the post-transfection LAV F17 vaccine Mode of administration: subcutaneously into the upper-outer triceps/deltoid area of the subject's arm; vaccination will be given in the non-dominant arm whenever possible Schedule Varied, 2 vaccinations per volunteer in a heterologous prime-boost strategy. First dose on Day 0 (PIV) AND a second dose (LAV) on Day 180 for group 1. First dose on Day 0 (PIV) AND a second dose (LAV) on Day 90 for group 2.

This study is intended to further evaluate the safety and reactogenicity of 2 tetravalent dengue vaccine (TDENV) candidates administered in a heterologous prime boost fashion with PIV followed by LAV 180 days later and to evaluate the safety and reactogenicity of a previously untested vaccination schedule consisting of PIV followed by LAV 90 days later.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 42 years of age (inclusive) at the time of consent
* Able to provide written informed consent
* Healthy as established by medical history and clinical examination and basic hematologic laboratory analysis before entering into the study
* Able and willing to comply with the requirements of the protocol (eg, document events in memory aid, return for follow-up visits, etc.)
* Dengue exposure naïve as established by pre-enrollment dengue PRNT testing and questioning of volunteer
* Female subject of non-childbearing potential (non-childbearing potential is defined as having either a current bilateral tubal ligation at least 3 months prior to enrollment or a history of an hysterectomy, bilateral oophorectomy, or is post-menopause(12 months or more since last menstrual period)) or Female subject of childbearing potential may be enrolled in the study, if the subject has:

  * Practiced adequate contraception for 30 days prior to vaccinations, and
  * A negative urine pregnancy test on each day of vaccination, and
  * Agreed to continue adequate contraception through at least 3 months following last vaccination

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine or device) other than the study vaccines during the period starting 30 days preceding the first dose of study vaccine and/or planned use during the study period
* Chronic administration (defined as more than 14 days in total) of prescription immunosuppressants or other prescription immune-modifying drugs during the period starting 180 days prior to the first vaccine dose

  * For corticosteroids, this will mean prednisone ≥ 20 mg/d or equivalent
  * Inhaled and topical steroids are allowed
* History of or active use of cancer chemotherapy or radiation therapy for the treatment of cancer
* Receipt or planned receipt of a vaccine/product outside the study protocol within 30 days of each scheduled dose of an investigational product
* Planned administration of any flavivirus vaccine, to include licensed vaccines for Yellow Fever or Japanese Encephalitis Virus as well as other investigational vaccines for dengue, Zika, West Nile, other flavivirus, for the entire study duration
* Previous receipt of a foreign or investigational dengue vaccine
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device)
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of, or current, auto-immune disease
* History of any reaction or hypersensitivity likely to be triggered by any component of the vaccines or related to a study procedure (This includes hypersensitivity reactions to alum, streptomycin, neomycin, or any other flavivirus vaccine, such as Yellow Fever virus and Japanese Encephalitis virus vaccines)
* Major congenital defects or serious chronic illness
* History of any chronic neurological disorders or chronic and/or uncontrolled seizures
* Acute infectious disease and/or fever (oral body temperature ≥ 100.4°F/38.0°C) at the time of enrollment (a subject with a minor illness, ie, mild diarrhea, mild upper respiratory infection, etc., without fever, may be enrolled at the discretion of the investigator)
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by history, physical examination or laboratory screening tests
* Receipt of immunoglobulins or any blood products during the period starting 90 days preceding the first dose of study vaccine or planned receipt during the study period
* Donated blood within 8 weeks before first scheduled investigational vaccine receipt or planned donation of blood products throughout the study period
* History of chronic alcohol abuse and/or drug abuse that, in the opinion of the investigator, could result in poor compliance with study requirements.
* Pregnant or breastfeeding female or female planning to become pregnant or planning to discontinue contraceptive precautions
* A planned move to a location that will prohibit compliance with the requirements of the trial
* Subject seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV)
* Safety laboratory test results that are outside the acceptable values at screening:

  * > 110% upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, creatinine, serum urea nitrogen (SUN) and bilirubin (total and direct)
  * < 100% lower limit of normal (LLN) or > 120% ULN for hemoglobin, hematocrit and platelet count
  * < 75% LLN or >110% ULN for total white blood cell count (WBC) Note: Per guidance in section 8.1, abnormal lab(s) may be repeated x1 in the screening window provided the total amount of blood drawn for all screening labs does not exceed 50 mL.
* Active Diabetes or active peptic ulcer disease (PUD)
* Diagnosis with Bipolar Disorder or Schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition, which in the opinion of the investigator prevents the subject from meeting all requirements of the study
* Chronic migraine headaches, defined as more than 15 headache days per month over a 3 month period of which more than 8 are migrainous, in the absence of medication over use
* Chronic medical condition that, in the opinion of the investigator, impacts subject safety
* Any other condition which, in the opinion of the investigator, prevents the subject from meeting all requirements of the study.
* Do not wish to have their blood stored and used for future research

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects With At Least One Local Solicited Adverse Events (AE) during the 28 Day Follow-up After Prime and Boost Vaccinations | 28 day follow-up period
  The number of subjects with at least one local solicited adverse event (AE), at least one general solicited AE and any solicited AE during the 28-day follow-up period for prime and boost vaccination will be tabulated with 95% confidence interval (CI) after each vaccine dose and overall.

SECONDARY OUTCOMES:
Number of subjects reporting at least one of each type of unsolicited AE during the 28-day follow-up period after each vaccination | 28 day follow-up period
  The number of subjects reporting at least one of each type of unsolicited AE during the 28-day follow-up period after each vaccination will be tabulated with 95% CIs

OTHER OUTCOMES:
The proportion of subjects with at least one report of any SAE during the 28 day follow-up period after each vaccination | 28 day follow-up period
  The proportion of subjects with at least one report of any SAE and reported up to 28 days (Day 0-Day 27) after each vaccination will be tabulated with 95% CIs.
The proportion of subjects with abnormal hematological or biochemical laboratory values | Days 0, 7 and 28 after each vaccination
  The proportion of subjects with abnormal hematological or biochemical laboratory values will be presented with 95% CIs at baseline and at each specified time point.
Number of withdrawals due to potential immune-mediated diseases (pIMDs), SAEs and AEs during the entire study | up to 18 months
  Number of subject withdrawals due to potential immune-mediated diseases (pIMDs), SAEs and AEs during the entire study
GMTs of subjects with detectable dengue viremia | dailiy testing between days 6 and 14 after vaccination
  GMT of subjects with detectable dengue viremia measured in days after each vaccination
Microneutralizing (MN) and flow cytometry based neutralizing dengue antibody titers | Day 0, 28 days after, immediately prior to the second (boost) vaccination (90 or 180 days), then 28 days, 180 days, 270 days, and 360 days following the second(boost) vaccination
  Microneutralizing (MN) and flow cytometry based neutralizing dengue antibody titers before first (prime) vaccination, 28 days after, immediately prior to the second (boost) vaccination (90 or 180 days), then 28 days, 180 days, 270 days, and 360 days following the second(boost) vaccination.
GMTs of neutralizing antibody against each DENV serotype (1-4) | Day 0 and Day 28 after each immunization and immediately prior to the boost vaccination (day 90 or 180) for the prime vaccination and at Days 180, 270 and 360 following boost vaccination
  GMTs of neutralizing antibody against each DENV serotype (1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Simon D Pollett, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- WRAIR, Clinical Trials Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT03141138/Prot_000.pdf